CLINICAL TRIAL: NCT01041625
Title: An Open-Label Pilot Study to Evaluate the Safety and Efficacy of Apremilast (CC-10004) in the Treatment of Moderate to Severe Lichen Planus
Brief Title: Pilot Study of Apremilast (CC-10004) in the Treatment of Moderate to Severe Lichen Planus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Virginia Clinical Research, Inc. (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: David M. Pariser, MD, Virginia Clinical Research Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCR 001; 107047 (Other: FDA IND Number)
Record Dates: First submitted 2009-12-30; First posted 2010-01-01 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Lichen Planus
Keywords: Lichen Planus
MeSH Terms: conditions — Lichen Planus | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apremilast (Experimental): Apremilast 20 mg PO administered BID over 12 weeks
  Interventions: Drug: Apremilast (CC-10004)

INTERVENTIONS:
Drug: Apremilast (CC-10004) — Apremilast 20 mg tablet PO administered BID over 12 weeks
  Other Names: N-{2-[1-(3-ethoxy-4-methoxyphenyl)-2-(methylsulfonyl)ethyl]-1,3-dioxoisoindolin-4-yl}acetamide (S enantiomer)

SUMMARY:
This study is designed to demonstrate to efficacy and safety of Apremilast 20mg oral administration twice daily over 12 weeks in subjects with moderate to severe lichen planus. The hypothesis is that the subjects will achieve a significant clinical improvement in their skin disease according to a specialized physician grading scale.

DETAILED DESCRIPTION:
This is a phase 2, single center, non-randomized, open label efficacy and safety study designed to characterize the response of Apremilast 20 mg oral administered twice daily over 12 weeks in subjects with moderate to severe lichen planus. The hypothesis and ideal primary end point will be that subjects achieve significant clinical response in cutaneous disease defined as a 2 or more grade improvement of the physician global assessment (PGA) after 12 weeks of treatment.

Many various therapies have been used to treat LP including topical and oral corticosteroids, retinoids, cyclosporine, griseofulvin, dapsone and phototherapy, but often with disappointing response.4 It is an inflammatory condition whose pathogenesis involves damage to basal keratinocytes by alloreactive T cells through the release proinflammatory cytokines, such as TNF-α and IFN-γ.1 Significantly elevated levels of such inflammatory mediators are present in tissue from LP lesions compared to normal controls.5 Based on these observations, the investigation of Apremilast, due to its ability to inhibit multiple inflammatory cytokines, for the treatment of moderate to severe LP is warranted.

The primary objective of this study is to evaluate the clinical efficacy of Apremilast in subjects with moderate to severe lichen planus after 12 weeks of treatment. Other objectives are to evaluate the safety and tolerability of Apremilast, effects on quality of life, and efficacy for mucosal disease if present.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form
* Must be male or female and aged ≥ 18 years at time of consent
* Must be able to adhere to the study visit schedule and other protocol requirements
* Subjects must have stable cutaneous lichen planus appropriate for systemic therapy based on the following criteria:

  * Rated PGA of ≥ 3 (moderate or severe) AND
  * ≥ 20 distinct lesions of lichen planus OR
  * Refractory to topical corticosteroid therapy (at least 4 weeks of high potency corticosteroid without significant improvement) OR
  * Severe itching/pain that significantly impairs activities of daily living (i.e. working, school, sleep, etc.)
* Subjects using topical corticosteroids must be tapered and must undergo a washout period prior to initiation of the study. The washout period for topical corticosteroids is 2 weeks.
* Must meet the following laboratory criteria:

  * Hemoglobin > 12 g/dL
  * White blood cell (WBC) count ≥ 3000 /μL (≥ 3.0 X 109/L) and ≤ 14,000/μL (< 14 X 109/L)
  * Platelets ≥ 100,000 /μL (≥ 100 X 109/L)
  * Serum creatinine ≤ 1.5 mg/dL (or ≤ 133 μmol/L)
  * Total bilirubin ≤ 2.0 mg/dL
  * Aspartate transaminase (AST [serum glutamic oxaloacetic transaminase, SGOT]) and alanine transaminase (ALT [serum glutamate pyruvic transaminase, SGPT]) ≤ 1.5x upper limit of normal (ULN)
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening (Visit 1). In addition, sexually active FCBP must agree to use TWO of the following adequate forms of contraception while on study medication: oral, injectable, or implantable hormonal contraceptives; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner while on study. A FCBP must agree to have pregnancy tests every 4 weeks while on study.
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with FCBP while on study medication and for 84 days after taking the last dose of study medication

Exclusion Criteria:

* Inability to provide voluntary consent
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or breastfeeding
* Systemic fungal infection
* History of active mycobacterial infection with any species (including Mycobacterium tuberculosis) within 3 years prior to screening visit. Subjects with Mycobacterium tuberculosis infection more than 3 years prior to screening visit are allowed if successful treatment was completed at least 3 years prior to randomization and is documented and available for verification.
* Latent Mycobacterium tuberculosis infection as indicated by a positive Purified Protein Derivative [PPD] skin test. Subjects with a positive PPD skin test and documented completion of treatment for latent TB are eligible. Subjects with a positive PPD skin test and not treated or no documentation of completion of treatment are ineligible.
* If QuantiFERON® test is performed instead of the PPD test, only those with a negative QuantiFERON® test are allowed in the study.
* History of incompletely treated Mycobacterium tuberculosis infection as indicated by

  * Subject's medical records documenting incomplete treatment for Mycobacterium tuberculosis
  * Subject's self-reported history of incomplete treatment for Mycobacterium tuberculosis
* History of recurrent bacterial infection (at least 3 major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years)
* Clinically significant abnormality on the chest x-ray (CXR) at screening. Chest x-rays performed within 3 months prior to start of study drug are acceptable.
* Use of topical cyclosporine, tacrolimus, or pimecrolimus within 2 weeks prior to start of study drug
* Use of systemic or intralesional corticosteroids, systemic retinoids, antimalarials, azathioprine, methotrexate, mycophenolate mofetil, dapsone, thalidomide, sulfasalazine, cyclosporine, metronidazole, griseofulvin, or phototherapy within 4 weeks prior to start of study drug
* Use of etanercept within 8 weeks prior to start of study drug.
* Use of adalimumab or infliximab within 12 weeks prior to start of study drug
* Use of alefacept within 24 weeks prior to start of study drug.
* Use of any investigational medication within 4 weeks prior to start of study drug or 5 pharmacokinetic/pharmacodynamic half-lives (whichever is longer)
* Any clinically significant abnormality on 12-lead ECG at screening
* History of congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency [CVID])
* Hepatitis B surface antigen positive or Hepatitis B core antibody positive at screening
* History of Human Immunodeficiency Virus (HIV) infection
* Antibodies to Hepatitis C at screening
* Positive ANA at screening visit
* Malignancy or history of malignancy (except for treated [ie, cured] basal- cell skin carcinomas > 3 years prior to screening)
* Presence of any other skin condition which may affect the evaluations of the study disease.
* Clinical picture suspicious for lichenoid drug eruption.
* Subjects whose lichen planus is predominantly hypertrophic, follicular, atrophic, or bullous variant.
* Lichen planus involving only mucosa or nails.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving significant clinical response in cutaneous disease defined as a 2 or more grade improvement of the physician global assessment (PGA) after 12 weeks of treatment. | 12 weeks

SECONDARY OUTCOMES:
Proportion of subjects with mucosal involvement who achieve a significant clinical response in mucosal disease defined as physician global assessment of mucosal disease (PGAMD) of "complete resolution" or "marked improvement" after 12 weeks of treatment. | 12 weeks
Change in the subjects' target area lesion count after 12 weeks of treatment relative to baseline. | 12 weeks
Change in the subjects' target area lesion severity score (TALSS) after 12 weeks of treatment relative to baseline. | 12 weeks
Proportion of subjects who achieve a subject global assessment of "complete resolution" or "marked improvement" after 12 weeks of treatment. | 12 weeks
Change in the subjects' dermatology life quality index (DLQI) score after 12 weeks of treatment relative to baseline. | 12 weeks
Change in the subjects' assessment of itching on a visual analogue scale (VAS) after 12 weeks of treatment relative to baseline. | 12 weeks
Safety and tolerability of Apremilast (type, frequency, severity, and relationship of adverse events to study treatment) | 16 weeks total (12 weeks treatment, 4 weeks observation)

CONTACTS AND LOCATIONS:
Overall Officials: David M Pariser, MD, Principal Investigator — Virginia Clinical Research, Inc.; Clare E Foss, MD, Study Chair — Eastern Virginia Medical School
Locations (1):
- Virginia Clinical Research Inc., Norfolk, Virginia, United States

REFERENCES:
- [Background] Boyd AS, Neldner KH. Lichen planus. J Am Acad Dermatol. 1991 Oct;25(4):593-619. doi: 10.1016/0190-9622(91)70241-s. PMID 1791218
- [Background] Silverman S Jr, Gorsky M, Lozada-Nur F, Giannotti K. A prospective study of findings and management in 214 patients with oral lichen planus. Oral Surg Oral Med Oral Pathol. 1991 Dec;72(6):665-70. doi: 10.1016/0030-4220(91)90007-y. PMID 1812447
- [Background] Cribier B, Frances C, Chosidow O. Treatment of lichen planus. An evidence-based medicine analysis of efficacy. Arch Dermatol. 1998 Dec;134(12):1521-30. doi: 10.1001/archderm.134.12.1521. PMID 9875189
- [Background] Chen X, Liu Z, Yue Q. The expression of TNF-alpha and ICAM-1 in lesions of lichen planus and its implication. J Huazhong Univ Sci Technolog Med Sci. 2007 Dec;27(6):739-41. doi: 10.1007/s11596-007-0632-x. PMID 18231758
- [Background] Bolognia JL, Jorizzo JL, Rapini RP. Dermatology. 2nd ed. Philadelphia, Pa: Elsevier: 2008.
- [Derived] Paul J, Foss CE, Hirano SA, Cunningham TD, Pariser DM. An open-label pilot study of apremilast for the treatment of moderate to severe lichen planus: a case series. J Am Acad Dermatol. 2013 Feb;68(2):255-61. doi: 10.1016/j.jaad.2012.07.014. Epub 2012 Aug 19. PMID 22910104